CLINICAL TRIAL: NCT00143299
Title: A 52-Week, Double-Blind, Placebo-Controlled, Randomized, Multicenter Study Evaluating the Safety of Varenicline Tartrate ( CP-526,555) for Smoking Cessation
Brief Title: A 52-Week Placebo-Controlled Study Evaluating the Safety of Varenicline
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051037
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2007-06-04 (Estimated); Status verified 2007-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

INTERVENTIONS:
Drug: varenicline (CP-526,555)

SUMMARY:
The primary purpose of this study is to obtain safety information on cigarette smokers treated with 52 weeks of varenicline regardless of smoking status.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have smoked an average of at least 10 cigarettes per day during the past year and over the month prior to the screening visit, with no period of abstinence greater than 3 months in the past year.

Exclusion Criteria:

* Subjects with clinically significant, recent cardiovascular disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375
Dates: Start 2003-10; Study Completion 2005-03

PRIMARY OUTCOMES:
Summarization of safety data in smokers treated with either varenicline or placebo.

SECONDARY OUTCOMES:
Information will be collected for the 7 day point prevalence of smoking cessation.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (8):
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Harleysville, Pennsylvania
  - Pfizer Investigational Site, Richmond, Virginia
- Pfizer Investigational Site, Woodville South, South Australia, Australia

REFERENCES:
- [Derived] Williams KE, Reeves KR, Billing CB Jr, Pennington AM, Gong J. A double-blind study evaluating the long-term safety of varenicline for smoking cessation. Curr Med Res Opin. 2007 Apr;23(4):793-801. doi: 10.1185/030079907x182185. PMID 17407636